CLINICAL TRIAL: NCT06835374
Title: Comparative Assessment of Reflux Esophagitis in Cases With and Without Esophageal Motility Disorders
Brief Title: Comparative Assessment of Esophagitis in Cases With and Without Esophageal Motility Disorders: A Prospective Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director, Asian Institute of Gastroenterology, India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REP
Record Dates: First submitted 2025-02-08; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assesment of reflux esophagitis in cases with esophageal motility (Active Comparator): Reflux esophagitis can be found in Endoscopy report.
  Interventions: Procedure: Per oral endoscopy myotomy (Per oral endoscopy myotomy)
- Assesment of reflux esophagitis in cases without esophageal motility (Placebo Comparator): Reflux esophagitis can be found in cases in normal gastroesophageal reflux disease condition patients
  Interventions: Procedure: Endoscopy procedure

INTERVENTIONS:
Procedure: Per oral endoscopy myotomy (Per oral endoscopy myotomy) — POEM is the procedure to reduce the symptoms of dysphagia, regurgitation.
  Arms: Assesment of reflux esophagitis in cases with esophageal motility
Procedure: Endoscopy procedure — Endoscopy procedure is required to rule out type of reflux disease
  Arms: Assesment of reflux esophagitis in cases without esophageal motility

SUMMARY:
Achalasia is a neuro-degenerative disorder marked by changes in the peristalsis of the esophagus and the lack of relaxation in the lower esophageal sphincter (LES), thought to be due to damage to the myenteric plexus with an unknown cause.1 Per-oral endoscopic myotomy (POEM) is an established endoscopic treatment modality for achalasia. Leading gastrointestinal (GI) societies endorse POEM as one of the primary treatment option for achalasia.This study aims to characterize and compare the morphological characteristics of reflux related erosions after the POEM procedures versus those in cases without esophageal motility disorders.

Data collection

1. Demographic characteristics: Age, gender, type of achalasia
2. Manometry findings (pre and post POEM): integrated relaxation pressure, lower esophageal sphincter pressure
3. Comorbidities
4. Medications
5. Eckardt score: before procedure and 3-months after Procedure
6. POEM procedure details: length of esophageal and gastric myotomy, adverse events, length of hospital stay
7. Evaluation at 3-months Symptom: standardized questionnaire (GERDQ) Endoscopy: grade of esophagitis Erosions vs ulcers Dimension of erosions Anatomical location (according to clock)

DETAILED DESCRIPTION:
POEM will be performed using a standardized technique.8 The patients will be prescribed a single dose anti-secretory medicine (equivalent to 40 mg esomeprazole) for two months after POEM. Consecutive patients who meet the inclusion and exclusion criteria will be followed up after 3 months. PPIs will be discontinued for at least 4 weeks prior to objective evaluation of GERD. Each patient returning after 3 months for follow up will undergo several follow up examinations, including GERD questionnaire scoring, Esophagogastroduodenoscopy, 24 hour pH impedance test. Presence of endoscopically visible esophagitis . Endoscopic findings such as anatomical location, dimensions of the mucosal breaks will be compared to general population with diagnosis of GERD who have endoscopically visible esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18y,
2. confirmed diagnosis of Achalasia,
3. No contraindication to POEM,
4. erosive esophagitis on endoscopy

Exclusion Criteria:

1. Non-esophageal esophageal motility disorders,
2. Treatment other than POEM,
3. current PPI use before assessment for GERD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
comparison of reflux esophagitis in cases who undergo POEM procedure versus those without esophageal motility disorders | 3 months
  Reflux esophagitis can be calculated as grade B category (red colour scar found in esophagus mucosa) during endoscopy procedure
Assessment of the , esophageal acid exposure | 6 months
  esophageal acid exposure is a value indicates higher reflux can be calculated in ph impedence report

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Nabi Dr Mohammed, MBBS MD, Principal Investigator — AIG Hospitals; Chinmay Dr Hegde, MBBS MD, Principal Investigator — AIG Hospitals
Locations (1):
- Asian Institute of Gastroenterology Hospital, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No